CLINICAL TRIAL: NCT04117217
Title: Analysis of Laboratory Markers to Predict Risk of Catheter Related Thrombosis
Brief Title: Risk Factors for Thrombosis in Children With Central Venous Lines
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Other Study IDs: 1701146088R002
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2019-10

CONDITIONS: Pediatric Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Central venous lines: Patients having a central venous catheter placed at Banner University Medical Center, University of Arizona
  Interventions: Diagnostic Test: Labs drawn
- Cardiac catheterization: Patients undergoing a cardiac catheterization procedure done at Banner University Medical Center, University of Arizona
  Interventions: Diagnostic Test: Labs drawn

INTERVENTIONS:
Diagnostic Test: Labs drawn — We will collect blood samples/biomarkers at the time of enrollment.

SUMMARY:
This project addresses the role of lab markers around the time of central line placement in predicting risk of thrombosis in pediatric patients with central venous lines being placed. The project proposes an innovative way to predict higher risk of thrombosis in the pediatric population to give clinicians a valid tool to guide clinical practice for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 5 kg and less than 18 years of age.
* Patients having a central venous catheter or cardiac catheterization performed

Exclusion Criteria:

* prior history of thrombosis
* patients with hemophilia A or B

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients having central venous line placement
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Thrombosis | within one year of enrollment
  Patients will be enrolled during the time of central line placements and labs would be drawn during line placement. Patients will be followed prospectively for a catheter related t thrombosis event or not. Lab markers and clinical states of patients who develop or do not develop a thrombosis will be analyzed

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No